CLINICAL TRIAL: NCT02183493
Title: Relative Bioavailability of a 5 mg BI 1356 Tablet Administered With and Without Food to Healthy Male and Female Subjects in an Open, Randomised, Single Dose, Two-way Crossover, Phase I Trial
Brief Title: Bioavailability of BI 1356 Administered With and Without Food to Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1218.34
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin

ARMS (2):
- Fed administration of BI 1356 (Experimental)
  Interventions: Drug: BI 1356
- Fasted administration of BI 1356 (Active Comparator)
  Interventions: Drug: BI 1356

INTERVENTIONS:
Drug: BI 1356

SUMMARY:
To investigate the food effect on the relative bioavailability and pharmacokinetics of a 5 mg BI 1356 tablet administered as a single dose

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria:

  -- Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
* Age ≥ 18 and Age ≤ 50 years
* BMI ≥ 18.5 and BMI ≤ 29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination deviating from normal and of clinical relevance. Repeated measurement of a systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs within one month or less than 10 half-lives of the respective drug prior to first study drug administration and during the trial except if a relevant interaction can be ruled out
* Participation in another trial with an investigational drug within two months prior to first study drug administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (average consumption of more than 20 g/day in females and 30 g/day in males)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to the start of study)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for torsades de points (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

For female subjects:

* Positive pregnancy test, pregnancy or planning to become pregnant during the study or within 2 months after study completion
* No adequate contraception during the study and until 2 months after study completion, i.e. not any of the following: implants, injectables, combined oral contraceptives, intrauterine device (IUD) , sexual abstinence for at least 1 month prior to enrolment, vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (including hysterectomy). Females, who do not have a vasectomised partner, are not sexually abstinent or surgically sterile will be asked to use an additional barrier method (e.g. condom, diaphragm with spermicide)
* Lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of BI 1356 in plasma over the time interval from 0 to 72 h (AUC0-72) | up to 72 hours after start of treatment
Maximum measured concentration (Cmax) of BI 1356 in plasma | up to 96 hours after start of treatment

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 1356 in plasma at different time points | up to 96 hours after start of treatment
Time from dosing to the maximum concentration (tmax) of BI 1356 in plasma | up to 96 hours after start of treatment
Terminal elimination rate constant (λz) in plasma | up to 96 hours after start of treatment
Terminal half-life (t1/2) of BI 1356 in plasma | up to 96 hours after start of treatment
Mean residence time of BI 1356 in the body after oral administration (MRTpo) | up to 96 hours after start of treatment
Apparent clearance of BI 1356 in the plasma after extravascular administration (CL/F) | up to 96 hours after start of treatment
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) | up to 96 hours after start of treatment
Number of patients with adverse events | up to 11 weeks
Assessment of tolerability on a 4-point scale by investigator | 14 days after last study drug administration